CLINICAL TRIAL: NCT05187533
Title: Efficacy of the Sphenopalatine Ganglion Stimulation Osteopathic Protocol in Patients with Ocular and Oral Dryness
Brief Title: Sphenopalatine Ganglion Stimulation for Ocular and Oral Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOBA-2021-23
Record Dates: First submitted 2021-10-28; First posted 2022-01-12 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease; Xerostomia
Keywords: dry eye disease; dryness; osteopathy; Keratoconjunctivitis sicca; Saliva cytokines; Saliva-producing glands; Sjögren´s syndrome; Sphenopalatine ganglion; Tear-producing glands; Tear cytokines; Tear film; Xerostomia
MeSH Terms: conditions — Dry Eye Syndromes; Xerostomia; Keratoconjunctivitis Sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild dry eye disease (Other): Osteopathic protocol of sphenopalatine ganglion stimulation
  Interventions: Other: Osteopathic protocol of Sphenopalatine Ganglion Stimulation
- Moderate dry eye disease (Other): Osteopathic protocol of sphenopalatine ganglion stimulation
  Interventions: Other: Osteopathic protocol of Sphenopalatine Ganglion Stimulation
- Severe dry eye disease (Other): Osteopathic protocol of sphenopalatine ganglion stimulation
  Interventions: Other: Osteopathic protocol of Sphenopalatine Ganglion Stimulation

INTERVENTIONS:
Other: Osteopathic protocol of Sphenopalatine Ganglion Stimulation — Sphenopalatine Ganglion Stimulation to improve lacrimal and salivary gland secretion to improve ocular and oral dryness

SUMMARY:
Dry Eye Disease (DED) is a multifactorial pathology characterized by inflammation of the lacrimal functional unit that develops in ocular surface pathology, severely affecting patients quality of life. The core of the treatment relies at present in antinflammatory topical therapies, which are still scarce.

The investigators hypothesize that osteopathy-based techniques may help these patients by influencing the central involvement regarding parasympathetic innervation of tear and saliva-secreting glands.

The aim of this osteopathic treatment protocol is to release the involved structures in the tear-secreting system innervation, such as the sphenopalatine ganglion. In addition, this ganglion innervates the minor salivary glands, therefore it is intended to help patients suffering from xerostomia.

The hypothesis then is that a systemic protocol treatment can help balance both parts of the vegetative nervous system (sympathetic and parasympathetic) with the objective of increasing the secretion of tear and saliva in patients with ocular and oral dryness (DED and xerostomia, respectively), thus improving their clinical situation.

This osteopathic protocol does not have the potential to cause adverse effects. The main objective is to analyze the efficacy of this protocol application in terms of improving symptoms and signs of ocular and oral dryness, tear film quality and inflammation molecule levels in tears and saliva.

DETAILED DESCRIPTION:
This clinical study intended to offer an alternative therapeutic tool for a disease, dry eye, that is highly prevalent, causes a decreased in the quality of life and work productivity, and whose pharmacologic treatment is very limited.

The osteopathy protocol consists of an initial assessment of the cranial vault and 7 techniques through which the different structures involved are treated and are as follows: 1) balance of the cranio-sacral system; 2) reharmonization of sphenobasilar synchondrosis; 3) and 4) release of the bony components in the pterygo-palatine fossa (maxillas and sphenoid); 5) and 6) release of the bony components in relation with the main lacrimal gland (frontal and front-malar suture); and 7) sphenopalatine ganglion stimulation. The patient is always in supine position and the investigator is standing on the side.

The proposed osteopathy protocol is innocuous, with no possible adverse effects. The main objective is to analyze the efficacy of this protocol application in terms of improving symptoms and signs of ocular and oral dryness, tear film quality and inflammation molecule levels in tears and saliva.

Recruited patients will have dry eye disease (and subsequently ocular dryness) and oral dryness (xerostomia). Inclusion/exclusion criteria are detailed in the corresponding section below, as well as all outcome measures.

All COVID19-related sanitary regulations will be strictly followed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old.
* Patients diagnosed with Dry eye disease (DED) and suffering symptoms of ocular and oral dryness for at least 6 months.
* "Dry eye" symptoms must have a score of > 2 (0-4 range) in mSIDEQ questionnaire.
* Ocularly symptomatic patients (OSDI > 12) despite the medication, medical devices and/or therapeutic measures carried out until the inclusion.
* Symptomatic patients in terms of oral dryness (XI-Sp > 11) despite the medication, medical devices and/or therapeutic measures carried out until the inclusion.
* Schirmer I test, without topical anesthesia, must have an initial value of ≥ 1 mm and <10 mm.
* Not included in any other clinical pharmacological trial or study (medical devices are excluded) in the last 3 months.
* Signed informed consent and ability to complete all study visits.

Exclusion Criteria:

* Irreversible anatomical alteration of the lacrimal glands (watery, sebaceous or mucinic) or salivary, surgeries or by healing processes that affect eyelids and/or conjunctiva.
* Alteration in the autonomic nervous system.
* Another active ocular surface disease different from that caused by DED.
* Oral diseases, inflammations or acute injuries in the mouth (trauma, surgical intervention, etc.) in the last month or healing processes of the oral mucosa.
* Use of cyclosporine or topical tacrolimus started within < 3 months and/or steroids or blood derivatives started within < 1 month and that will not be maintained during the study.
* Use of orally drugs with exocrine hyposecretory side effects or that may affect the parasympathetic nervous system, unless the dose is stable during the previous month to inclusion and whose dose is not expected to vary throughout this study.
* Patients may be using any other medication, topical or systemic, unless the dose are the same for the duration of the study.
* Patients may be using artificial tears, moisturizers in general or blood derivatives, unless the dose was the same in the last month and has to be maintained at the same dose for the duration of the study.
* To have had any "in-office" method to manage DED or Meibomian gland dysfunction (pulsed light, thermal massages, etc.) in the last 6 months.
* Occlusion of the lacrimal puncta in the last month.
* Local (in cranial sphere) or general anesthesia in the last 3 months.
* Use of contact lenses, unless they stop using them for at least one week before inclusion and one week before each visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 6 Weeks
  Score value 0-48, where higher score means a worse outcome.
Ocular Surface Disease Index (OSDI) | 18 Weeks
  Score value 0-48, where higher score means a worse outcome.
Modified Single-Item Score Dry Eye-Questionnaire (mSIDEQ) | 6 Weeks
  Score value 0-28, where higher score means a worse outcome
Modified Single-Item Score Dry Eye-Questionnaire (mSIDEQ) | 18 Weeks
  Score value 0-28, where higher score means a worse outcome
Visual analogue Scale (VAS) | 6 Weeks
  Unique measurements 0-10, where higher score means a worse outcome
Visual analogue Scale (VAS) | 18 Weeks
  Unique measurements 0-10, where higher score means a worse outcome
Change in Dry Eye Symptoms Questionnaire (CDES-Q) | 6 Weeks
  First question compares how the patient is at the moment compared with last session in terms of "Equal", "Better" or "Worse". If better or worse is chose, two more questions measure how much improvement or worsening from a 0-10 scale, where higher score means a worse outcome.
Change in Dry Eye Symptoms Questionnaire (CDES-Q) | 18 Weeks
  First question compares how the patient is at the moment compared with last session in terms of "Equal", "Better" or "Worse". If better or worse is chose, two more questions measure how much improvement or worsening from a 0-10 scale, where higher score means a worse outcome.
Statistically significant amelioration in oral symptoms | 6 Weeks
  Enhancement in Xerostomia Inventory Spanish version (XI-Sp) test score 0-11, where higher score means a worse outcome.
Statistically significant amelioration in oral symptoms | 18 Weeks
  Enhancement in Xerostomia Inventory Spanish version (XI-Sp) test score 0-11, where higher score means a worse outcome.
Statistically significant improvement in tear secretion | 6 Weeks
  Schirmer I test, which test score is 0-35 mm, where lower score means a worse outcome.
Statistically significant improvement in tear secretion | 18 Weeks
  Schirmer I test, which test score is 0-35 mm, where lower score means a worse outcome.
Statistically significant improvement in salivary discharge | 6 Weeks
  Salivary flow rate, where flow rate below 0,1ml flow is considered hyposalivation.
Statistically significant improvement in salivary discharge | 18 Weeks
  Salivary flow rate, where flow rate below 0,1ml flow is considered hyposalivation.

SECONDARY OUTCOMES:
Decrease in tear collection time | 18 Weeks
  Statistically significant improvement in tear collection time, using a microcapillar of 1μl.
Increased salivary flow rate | 18 Weeks
  Statistically significant increased salivary flow rate, using Modified Fox Sreebny Technique.
Lipiflow interferometry - lipid layer thickness | 18 Weeks
  Statistically significant improvement in lipid layer thickness using Interferometry with Lipiview.
Lipiflow interferometry - incomplete blink rate | 18 Weeks
  Statistically significant improvement in incomplete blink rate using Interferometry with Lipiview.
Lipiflow interferometry - c-factor | 18 Weeks
  Statistically significant improvement in c-factor, using Interferometry with Lipiview.
Enhancement in Break-Up Time Test | 18 Weeks
  Statistically significant enhancement in Break-Up Time Test (normal >7 seconds) where lower score means a worse outcome.
Corneal Staining | 18 Weeks
  Statistically significant enhancement in Corneal Staining, using Oxford Scale and Cornea and Contact Lens Research Unit (CCLRU) Scale, score 0-5 where higher scores means worse outcome.
Significant beneficial change in molecules evaluated in tear or saliva | 18 Weeks
  The following putative salivary indicators of pain are assayed by enzyme-linked immunosorbent assay (ELISA): Cortisol (DRG Salivary Cortisol ELISA (DRG Instruments GmbH, Marburg, Germany), testosterone (DRG Instruments GmbH), sTNFαRII (Quantikine, Human sTNF RII/TNFRSF1B Immunoassay, R&D Systems, Minneapolis, MN, USA). sAA is

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No